CLINICAL TRIAL: NCT04039165
Title: Developing a Positive Psychology Intervention to Promote Health Behaviors in Metabolic Syndrome: A Randomized Controlled Pilot Trial
Brief Title: Developing a Positive Psychology Intervention to Promote Health Behaviors in Metabolic Syndrome: RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Rachel Millstein, Assistant Professor, Department of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019P001300
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: A group of participants, who will be randomized to wait-list control group, is assigned to a waiting list and receives intervention after the active treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will complete an 8-week group physical activity and positive psychology program, in which they will complete exercises related to increasing positive emotions and physical activity during and between the group sessions. They will track their activity (steps) and set personalized physical activity goals each week, and complete a group walk or indoor exercise during the group sessions. The investigators will ask questions about participants' health and health behaviors, and ask them to wear a physical activity monitor at the beginning and end of the program. During times when in-person visits cannot happen (e.g., COVID-19), we will do virtual group sessions instead of meeting at the clinics, conducted via videoconference platform (i.e., Zoom), the group walks will not happen, and all exercise will be done individually to comply with social distancing measures.
  Interventions: Behavioral: PP-MI Intervention
- Wait-list Control Comparison Group (No Intervention): Participants in the waitlist control group will not receive any active intervention during the initial study period (weeks 1-9). At Week 10, this group will receive the same intervention and assessments as described in the active treatment group above.

INTERVENTIONS:
Behavioral: PP-MI Intervention — The positive psychology exercises include gratitude-based activities, strengths-based activities, and meaning-based activities. The physical activity goal setting exercises include the following topics: health benefits, social resources, and neighborhood walkability.
  Arms: Intervention Group

SUMMARY:
Specific Aim #1 (Feasibility; primary aim): To assess the feasibility of the PP-MI group-based physical activity intervention and outcome assessments in patients with MetS.

Hypothesis: The PP exercises and MI-based goal-setting sessions will be feasible: most (≥50%) of participants will complete 6/9 exercises/sessions. Furthermore, the investigators will be able to obtain objective physical activity measurement follow-up data from at least 80% of enrolled participants at the end of the intervention and 24 weeks later.

Specific Aim #2 (Acceptability): To assess whether the intervention is acceptable to participants, as measured by ratings provided after each PP-MI session.

Hypothesis: The intervention will be acceptable: participants will rate the PP-MI exercises with a mean score of at least 7 out of 10 on ease of completion and helpfulness.

Specific Aim #3 (Outcomes): To assess whether this preliminary intervention appears to result in improvement of physical activity, related health behaviors (sedentary time, diet quality), psychological well-being (optimism, positive affect, anxiety, depression), and the exploratory outcomes of MetS-relevant physiological markers (e.g., blood pressure, weight, chart-reviewed lipids and HbA1C).

Hypothesis a: The intervention will lead to improvements in physical activity, related health behaviors, optimism and positive affect, reductions in depression and anxiety at 9 weeks and 24 weeks compared to baseline (or the start of the intervention, for the WLC group).

Hypothesis b: The hypothesis is that there will be improvements in the exploratory outcomes of the physiological markers, even if they do not reach significance.

DETAILED DESCRIPTION:
This randomized pilot trial will test a group-based PP-MI intervention adapted for patients with MetS. MGH outpatient community clinics will serve as the sources of recruitment and the sites of the groups. The investigators will recruit up to 64 patients with MetS to complete the study and provide follow-up data.

Baseline information about enrolled participants will be obtained from the patients, care providers, and the electronic medical record as required for characterization of the population. This information will include medical data related to MetS (e.g., blood sugar, blood pressure, body mass index, triglycerides, cholesterol), current medications, and sociodemographic data (age, gender, race/ethnicity, education, marital status).

Participants will attend 90-minute groups sessions that will be held at the clinics (MGH Healthcare Centers). The overall structure of each session will be: 30 minutes for positive psychology exercise review/discussion, 30 minutes for physical activity goal setting, education, and discussion, and 30 minutes for a group walk or indoor exercises in inclement weather. During times when in-person visits cannot happen (e.g., COVID-19), we will do virtual group sessions instead of meeting at the clinics, conducted via videoconference platform (i.e., Zoom). This study has been IRB-approved for waiver of informed consent documentation, so we will receive informed consent from our potential participants via verbal consent. We will mail/e-mail an IRB-approved study information fact sheet, providing them written details about our study before obtaining verbal informed consent. Each participant's verbal consent will be documented in REDCap. In addition, the group walks will not happen in these particular circumstances, and all exercise will be done individually to comply with social distancing measures.

Participants will be either randomized to an immediate intervention group or a wait-list control (WLC) group. The wait-list control group will start the intervention at Week 10, after the immediate intervention group completes its final session. Both groups will be asked to wear an Actigraph GT3x+ accelerometer for 1 week at baseline, then week 9, and week 24 for the intervention group, and at baseline, weeks 9, 17, and 33 for the WLC group. Accelerometers such as this one are considered to be the standard for measuring habitual physical activity. They are pedometer-size devices that attach to a belt and are worn at the waist. Participants will also be given a wrist-worn Fitbit to keep, which they will be asked to wear daily for the duration of the study in order to track their activity (steps).

Upon beginning the groups, participants will be provided with a treatment manual with weekly PP exercises, information about the importance of physical activity and related health behaviors, and how to set goals to improve these behaviors. The PI or a trained substitute will lead all groups.

For the first session, in the PP portion, participants will discuss and be assigned the first exercise- Gratitude for Positive Events- and will be instructed to complete the PP exercise during the next week. Prior to completing the exercise, participants will be asked to rate their current levels of happiness and optimism. Immediately after completing the exercise, participants will rate the ease of exercise completion, overall utility of the exercise, and their current levels of happiness and optimism, all using 10-point Likert scales. In the first goal-setting session, the investigators will discuss the importance of physical activity in MetS. Investigators will review instructions for Fitbit use and set a goal for monitoring their baseline physical activity over the next week. Fitbits will not be used as an outcome measure, but as a tool that participants can use to monitor their activity and set goals. Finally, the last 30 minutes will be spent doing a group walk around the local clinic neighborhood (or indoor exercise in the case of inclement weather). All group walks and exercises will be done at a pace comfortable for participants.

Participants will be asked to complete the 8 total weekly PP exercises, set physical activity goals, and attend as many group sessions as they can.

All sessions will include (a) a review and discussion of the past week's PP exercise, (b) a discussion of the rationale of the next week's PP exercise using the PP manual, and (c) assignment of the next week's PP exercise. For the goal-setting/MI portion, participants will (a) review their goals and steps from the prior week, (b) discuss techniques for improving physical activity (e.g., monitoring physical activity, taking standing breaks), and (c) set goals for the next week. The exercises and content for both PP and MI will be assigned in the same order for all participants receiving them.

At Weeks 9 and 24 (Weeks 17 and 33 for the wait-list control group), participants will complete the same self-report questionnaires that were administered at baseline. The investigators will collect the Actigraphs at baseline, weeks 9 and 24 (baseline, Weeks 9, 17 and 33 for the WLC group) and upload the data to assess for valid wear time. If participants have not worn them for enough time (>4 days), the investigators will send it home with them and ask them to re-wear it and mail it back.

ELIGIBILITY:
Inclusion Criteria:

Participants must have at least three of the five MetS criteria:

* Elevated abdominal obesity (waist circumference >102 cm in men or >88 cm in women)

  * If waist circumference is not available, body mass index (BMI) will be used as a surrogate measure based on prior research (BMI ≥29.1 kg/m2 for men and 27.2 kg/m2 for women).
* Elevated blood pressure (systolic ≥130 and/or diastolic ≥85 mm Hg or be on blood pressure medication).
* Serum triglycerides ≥150 mg/dL
* High-density lipoprotein (HDL) cholesterol <40 mg/dL in men or <50 mg/dL in women
* Fasting plasma glucose >100mg/dL.

OR

* Fewer than 3 MetS criteria but with PCP approval
* Suboptimal physical activity defined as ≤150 minutes/week moderate intensity activity, which represents less than national-level recommendations.

Exclusion Criteria:

* Inability to speak/read English
* Cognitive deficits impeding ability to participate or provide informed consent (measured by a 6-item screen)
* Illness likely to lead to death in the next 6 months per PCP
* Current treatment for cancer, liver, or renal disease
* Pregnancy
* Documented severe mental illness (e.g., psychosis, suicidality)
* No telephone access
* Inability to be physically active
* Diabetes or known or suggested cardiac disease, given that this is a primary prevention study.
* Participation in any other research studies or clinical trials that focus on increasing physical activities

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-07-25 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2023-01-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the PP-MI-Based Health Behavior Intervention | 8 weeks of group sessions
  Feasibility will be measured by examining the number of completed exercises.

SECONDARY OUTCOMES:
Acceptability of Intervention | 8 weeks
  Participants will rate the ease and usefulness of each weekly activity (0-10).
Physical Activity Adherence (Actigraph) | Baseline, weeks 9, 24 (baseline, weeks 9, 17, 33 for the WLC group)
  ActiGraph GT3X+ accelerometers are validated as measures of physical activity and have been used in numerous studies of physical activity in patients with medical illness. In this trial, participants will wear the accelerometer to assess the feasibility of doing so and to ensure adequate capture of physical activity.
Feasibility of Actigraph | Baseline, weeks 9, 24 (baseline, weeks 9, 17, 33 for the WLC group)
  Feasibility will be measured by examining the rates of use of the Actigraph.
Changes in Life Orientation Test- Revised Scores | Baseline, weeks 9, 24 (Baseline, weeks 17 and 33 for the WLC group)
  The LOT-R is a well-validated 6-item instrument used to measure dispositional optimism. (Range: 5-30)
Changes in Positive and Negative Affect Schedule Scores | Baseline, weeks 9, 24 (Baseline, weeks 17 and 33 for the WLC group)
  The positive affect items on the Positive and Negative Affect Schedule (PANAS), a well-validated scale used in other intervention trials, will be used to measure positive affect. (Range: 10-50)
Changes in The Hospital Anxiety and Depression Scale Scores | Baseline, weeks 9, 24 (Baseline, weeks 17 and 33 for the WLC group)
  The HADS will be used to measure depression and anxiety. This is a well-validated scale with few somatic symptom items that can confound mood/anxiety assessment in medically-ill patients. (Range: HADS-A, HADS-D; 0-21 each)
Changes in Barriers to Being Active Quiz Scores | Baseline, weeks 9, 24 (Baseline, weeks 17 and 33 for the WLC group)
  The BBAQ is a 21-item measure, published by the US Centers for Disease Control and Prevention (CDC), that explores seven main categories of barriers, including lack of time, energy, and resources. (Range: 0-63)
Changes in State Optimism Measure | Baseline, weeks 9, 24 (Baseline, weeks 17 and 33 for the WLC group)
  The SOM will be used to capture the changeable nature of optimism based on time and situation. (Range: 7-35)
Changes in The Medical Outcomes Study Short Form-12 Scores | Baseline, weeks 9, 24 (Baseline, weeks 17 and 33 for the WLC group)
  The SF-12 will be used to measure quality of life. This instrument has been used in many patient-oriented studies. (Range: SF-12 PCS and SF-12 MCS); range 0-100 each)
Changes in The International Physical Activity Questionnaire-Short Form Scores | Pre-baseline screening, weeks 9, 24 (Pre-baseline, weeks 17 and 33 for the WLC group)
  The IPAQ-SF is a validated scale that measures self-reported physical activity in the past 7 days in the domains of vigorous activity, moderate activity, and walking.
Changes in Behavioral Risk Factor Surveillance System Fruit and Vegetable Module | Baseline, weeks 9, 24 (Baseline, weeks 17 and 33 for the WLC group)
  The CDC's BRFSS Fruit and Vegetable Module is a brief questionnaire about frequency of eating different types of fruits and vegetables.
Changes in National Cancer Institute's Percentage Energy from Fat Screener Scores | Baseline, weeks 9, 24 (Baseline, weeks 17 and 33 for the WLC group)
  The National Cancer Institute's Percentage Energy from Fat Screen is a brief questionnaire that estimates people's typical percentage of energy derived from eating common fat-containing foods, as fat content is related to metabolic syndrome progression.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel A Millstein, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital- Revere Health Center, Revere, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No